CLINICAL TRIAL: NCT05535946
Title: A Randomized, Double-blind, Multicenter Phase III Study to Evaluate the Long-term Efficacy and Safety of ABX464 25 mg or 50 mg Once Daily as a Maintenance Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: ABTECT - Maintenance
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABX464-107
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ABX464

STUDY DESIGN:
Intervention Model Description: Among both induction studies, subjects assessed as responders will be randomized as follows into Part 1 of the maintenance study according to their induction treatment:
  * ABX464 Dose 50 mg QD
  * ABX464 Dose 25 mg QD
  * Placebo. All subjects with clinical response who were dosed with placebo in the induction studies will be randomized into the placebo group.
  Among both induction studies, subjects assessed as non-responders will be randomized as follows into Part 2 of the maintenance study according to their induction treatment:
  * ABX464 Dose 50 mg QD (all subjects who received 50 mg in induction)
  * ABX464 Dose 25 mg QD (all subjects who received 25 mg in induction)
  * Subjects who were allocated to placebo in the induction study will be randomized to obefazimod 50 mg or 25 mg in a blinded manner.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All eligible subjects will be randomized to either the double blind, placebo-controlled Part #1 (ABX464 50mg or 25mg or placebo) or randomized to double-blind Part #2 (ABX464 50mg or 25mg) depending on their clinical response at the end of induction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ABX464 50mg - Responder subjects at the end of induction (Placebo Comparator): Subjects will be orally dosed during 44 weeks
  Interventions: Drug: ABX464
- ABX464 25mg - Responder subjects at the end of induction (Placebo Comparator): Subjects will be orally dosed during 44 weeks
  Interventions: Drug: ABX464
- Placebo - Responder subjects at the end of induction (Placebo Comparator): Subjects will be orally dosed during 44 weeks
  Interventions: Drug: Placebo
- ABX464 50mg - Non responder subjects at the end of induction (Experimental): Subjects will be orally dosed during 44 weeks
  Interventions: Drug: ABX464
- ABX464 25mg - Non responder subjects at the end of induction (Experimental): Subjects will be orally dosed during 44 weeks
  Interventions: Drug: ABX464
- Long Term Extension (Experimental): At the end of the maintenance phase (week 44), subjects can continue their allocated treatment for up to 4 years. Once the maintenance phase is unblinded, subjects receiving placebo in the maintenance phase will be allocated to obefazimod 25 mg or can terminate the study.
  Interventions: Drug: ABX464

INTERVENTIONS:
Drug: ABX464 — Administered once daily, preferably in the morning, with food
  Other Names: Obefazimod
  Arms: ABX464 25mg - Non responder subjects at the end of induction; ABX464 25mg - Responder subjects at the end of induction; ABX464 50mg - Non responder subjects at the end of induction; ABX464 50mg - Responder subjects at the end of induction; Long Term Extension
Drug: Placebo — Administered once daily, preferably in the morning, with food
  Arms: Placebo - Responder subjects at the end of induction

SUMMARY:
This is a multicenter, randomized, placebo-controlled study to evaluate the long-term efficacy and safety of ABX464 50mg and 25mg administered once daily (QD) as maintenance therapy in subjects with moderately to severely active ulcerative colitis who have inadequate response, no response, a loss of response, or an intolerance to either conventional therapies [corticosteroids, immunosuppressant (i.e. azathioprine, 6-mercaptopurine, methotrexate)] and/or advanced therapies [biologics (TNF inhibitors, anti-integrins, anti-IL-23), and/or S1P receptor modulators, and/or JAK inhibitors].

This study is the maintenance phase of both previous induction studies ABX464-105 and ABX464-106.

DETAILED DESCRIPTION:
All eligible subjects who have completed either one of the induction studies above mentioned, will be given the opportunity to take part in the present ABX464-107 study which consists of 2 treatment phases.

This study consists of a 44-week maintenance treatment phase (Part 1 and Part 2), followed by a 4-year Long Term Extension (LTE) treatment phase and a 28-days follow-up period consisting in the End of Study (EOS) visit.

The maintenance phase is a 44-week double blind, placebo-controlled, phase. Subjects who are clinical responders after 8 weeks induction will be randomized to Part 1, and those who are non-clinical responders will be randomized to Part 2.

At the end of the 44-week maintenance phase, subjects will continue their allocated treatment until the maintenance phase is unblinded.

Once the study is unblinded, all subjects receiving obefazimod will continue their allocated treatment. Subjects receiving placebo will be allocated to obefazimod 25 mg or can terminate the study.

ELIGIBILITY:
Inclusion Criteria in maintenance phase:

* Subjects must have completed the induction treatment study (ABX464-105 or ABX464-106), and patients' clinical response status must be available.
* Subjects with a valid endoscopy performed at the end of the induction study and results from central reader available at Day 1.
* Subjects must understand, sign and date the written voluntary informed consent form at the visit prior to any protocol-specific procedures. For under-aged subjects, national requirements regarding consent should also be met.
* Women of childbearing potential (WOCBP) subjects and male subjects with WOCBP partner must agree to comply with contraception requirements as described in Section 4.4. (Contraception) of the protocol.
* Subjects must be able and willing to comply with study visits and procedures as per protocol.
* Subjects should be affiliated to a health insurance policy whenever required by a participating country or state

Inclusion criteria in LTE phase:

* Subject must have completed the maintenance phase
* Investigator and subject must assess and agree that the subject has received, and will continue to receive benefit from being in the study

Exclusion Criteria in maintenance phase:

* Subjects who permanently discontinued the study treatment during the induction study (either ABX464-105 or ABX464-106).
* Subjects who have developed any major illness/condition (eg. primary sclerosis cholangitis, Crohn's disease, colectomy, diverting ileostomy, colon cancer or colonic adenomas [low or high grade dysplasia]).
* Subjects with evidence of an unstable clinical condition (eg. toxic megacolon, fulminant colitis, bowel perforation, uncontrolled ischemic disease, congestive heart failure with NYHA class 3 or 4 symptoms) during the induction study that, in the investigator's judgment, will substantially increase the risk to the subject if he or she participates in the study.
* Subjects who plan to participate in other investigational studies during the maintenance study.
* Male or female planning a pregnancy, or pregnant female subjects
* Introduction during induction study of prohibited medications, dosages, surgical or non-medicinal procedures indicated for UC (except antidiarrheals and motility agents for acute diarrhea).
* Any changes in the laboratory values during the induction period that could jeopardize subject's safety in the opinion of the investigator. If any doubts, the investigator should contact the sponsor study medical monitor.
* Subject who is planning to receive live vaccine during the study.
* Subjects committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.

Exclusion criteria for LTE phase:

* Subject continues to satisfy exclusion criteria listed above for the maintenance phase
* Introduction during maintenance phase of prohibited medications, dosages, surgical or non-medicinal procedures indicated for UC (except antidiarrheals and motility agents for acute diarrhea).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects in clinical remission at Week 44 | Week 44
  The Part 1 primary objective is to compare the efficacy of ABX464 versus placebo on the proportion of subjects in clinical remission [SFS = 0 or 1, RBS = 0 and endoscopy sub-score = 0 or 1] at Week 44.
Number and percentage of all treatment-emergent adverse events (TEAEs) | Week 44
  The Part 2 primary objective is safety
Number and percentage of all serious adverse events (SAEs) | Week 44
  The Part 2 primary objective is safety
Number and percentage of all causally related TEAEs/SAEs | Week 44
  The Part 2 primary objective is safety

SECONDARY OUTCOMES:
Proportion of subjects with endoscopic improvement at Week 44 | Week 44
  To compare the efficacy of ABX464 versus placebo on endoscopic improvement (Mayo Endoscopic Subscore (MES) = 0 or 1) at Week 44
Proportion of subjects with corticosteroid-free clinical remission | Week 44
  To compare the efficacy of ABX464 versus placebo on corticosteroid-free clinical remission (clinical remission at Week 44 and corticosteroid free for at least 12 weeks prior to Week 44 in the subpopulation with corticosteroids at maintenance study entry)
Proportion of subjects with sustained clinical remission at Week 44 | Week 44
  To compare the efficacy of ABX464 versus placebo to sustain clinical remission at Week 44
Proportion of subjects with HEMI per Geboes scoring at Week 44 | Week 44
  To evaluate the efficacy of ABX464 on histologic-endoscopic mucosal improvement (HEMI) versus placebo at Week 44
Proportion of subjects with endoscopic remission at Week 44 | Week 44
  To compare the efficacy of ABX464 versus placebo on endoscopic remission (MES = 0) at Week 44
LTE Phase - Proportion of subjects in clinical remission at Year 1 | LTE Year 1
  To evaluate the efficacy of obefazimod on clinical remission [SFS = 0 or 1, RBS = 0 and endoscopy sub-score = 0 or 1] at Year 1
LTE Phase - Proportion of subjects in clinical remission at Year 4 | LTE Year 4
  To evaluate the efficacy of obefazimod on clinical remission [SFS = 0 or 1, RBS = 0 and endoscopy sub-score = 0 or 1] at Year 4
LTE Phase - Proportion of subjects with corticosteroid-free clinical remission in the subpopulation with corticosteroids at maintenance study entry | LTE Year 1
  To evaluate the efficacy of obefazimod on CS-free clinical remission (clinical remission at Year 1 and corticosteroid free for at least 12 weeks prior to Year 1 in the subpopulation with corticosteroids at maintenance study entry)
LTE Phase - Proportion of subjects with corticosteroid-free clinical remission in the subpopulation with corticosteroids at maintenance study entry) | LTE Year 4
  To evaluate the efficacy of obefazimod on CS-free clinical remission (clinical remission at Year 4 and corticosteroid free for at least 12 weeks prior to Year 4 in the subpopulation with corticosteroids at maintenance study entry)
LTE Phase - Proportion of subjects with endoscopic improvement at LTE Year 1 | LTE Year 1
  To evaluate the efficacy of obefazimod on endoscopic improvement (Mayo Endoscopic Subscore (MES) = 0 or 1)
LTE Phase - Proportion of subjects with endoscopic improvement at LTE Year 4 | LTE Year 4
  To evaluate the efficacy of obefazimod on endoscopic improvement (Mayo Endoscopic Subscore (MES) = 0 or 1)
LTE Phase - Proportion of subjects with endoscopic remission at LTE year 1 | LTE year 1
  To evaluate the efficacy of obefazimod on endoscopic remission ((Mayo Endoscopic Subscore (MES) = 0)
LTE Phase - Proportion of subjects with endoscopic remission at LTE year 4 | LTE year 4
  To evaluate the efficacy of obefazimod on endoscopic remission (Mayo Endoscopic Subscore (MES) = 0)
LTE Phase - Proportion of subjects with CS-free symptomatic remission by visit | 4 years
  To evaluate the efficacy of obefazimod on CS-free symptomatic remission (symptomatic remission (SFS = 0 or 1 and RBS = 0) and corticosteroid free for at least 12 weeks prior to Week 44 in the subpopulation with corticosteroids at maintenance study entry) by visit (every 3-month)
LTE Phase - Proportion of subjects with HEMI per Geboes scoring at LTE Year 1 | LTE Year 1
  To evaluate the efficacy of obefazimod on histologic endoscopic mucosal improvement (HEMI) per Geboes scoring
LTE Phase - Proportion of subjects with HEMI per Geboes scoring at LTE Year 4 | LTE Year 4
  To evaluate the efficacy of obefazimod on histologic endoscopic mucosal improvement (HEMI) per Geboes scoring
LTE Phase - Proportion of subjects with HEMR per Geboes scoring at LTE Year 1 | LTE Year 1
  To evaluate the efficacy of obefazimod on histologic endoscopic mucosal remission (HEMR) versus placebo
LTE Phase - Proportion of subjects with HEMR per Geboes scoring at LTE Year 4 | LTE Year 4
  To evaluate the efficacy of obefazimod on histologic endoscopic mucosal remission (HEMR) versus placebo
LTE Phase - Proportion of subjects with sustained clinical remission at LTE Year 1, in the sub-population of subjects with clinical remission at Week 44 | LTE Year 1
  To evaluate the efficacy of obefazimod on sustained clinical remission Sustained clinical remission for the LTE is defined as clinical remission assessed at an endoscopy visit during the LTE in the sub-population of subjects in clinical remission at Week 44.
LTE Phase - Proportion of subjects with sustained clinical remission at LTE year 4, in the sub-population of subjects with clinical remission at Week 44 | LTE year 4
  To evaluate the efficacy of obefazimod on sustained clinical remission Sustained clinical remission for the LTE is defined as clinical remission assessed at an endoscopy visit during the LTE in the sub-population of subjects in clinical remission at Week 44.
LTE Phase - Proportion of subjects with sustained endoscopic improvement at LTE Year 1, in the sub-population of subjects with endoscopic improvement at Week 44 | LTE Year 1
  To evaluate the efficacy of obefazimod on sustained endoscopic improvement
LTE Phase - Proportion of subjects with sustained endoscopic improvement at LTE Year 4, in the sub-population of subjects with endoscopic improvement at Week 44 | LTE year 4
  To evaluate the efficacy of obefazimod on sustained endoscopic improvement
LTE Phase - Proportion of subjects with symptomatic remission by visit | 4 years
  To evaluate the efficacy of obefazimod on symptomatic remission (SFS = 0 or 1 and RBS = 0) by visit (every 3-month)
LTE Phase - Proportion of subjects with sustained symptomatic remission by visit | 4 years
  To evaluate the efficacy of obefazimod on sustained symptomatic remission (SFS = 0 or 1 and RBS = 0) by visit (every 3-month), in the sub-population of subjects with symptomatic remission at Week 44
LTE Phase - Proportion of subjects with CS-free clinical remission at LTE Year 1 | LTE Year 1
  To evaluate the efficacy of obefazimod on CS-free clinical remission (clinical remission at Year 1 and CS-free for at least 12 weeks immediately prior to Year 1)
LTE Phase - Proportion of subjects with CS-free clinical remission at LTE Year 4 | LTE Year 4
  To evaluate the efficacy of obefazimod on CS-free clinical remission (clinical remission at Year 4 and CS-free for at least 12 weeks immediately prior to Year 4)

CONTACTS AND LOCATIONS:
Overall Officials: Severine Vermeire, MD, PhD, Principal Investigator — UZ Leuven, Belgium; Bruce Sands, MD, PhD, Principal Investigator — Mount Sinai Health System Digestive Disease Institute, New York USA
Locations (553):
- United States (137):
  - University of Alabama -Birmingham, Birmingham, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - Research Solutions of Arizona, PC, Litchfield Park, Arizona
  - Valleywise Health Medical Center, Phoenix, Arizona
  - GI Alliance, Sun City, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - National Institute of Clinical Research, Bakersfield, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Aurora Care Clinic, Costa Mesa, California
  - Citrus Valley Gastroenterology, Covina, California
  - University of California (San Diego), La Jolla, California
  - Gastro Care Institute, Lancaster, California
  - United Medical Doctors, Murrieta, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - California Medical Research Associates Inc., Northridge, California
  - Clinnova Research Solutions, Orange, California
  - Clinical Applications Laboratories, San Diego, California
  - Kaiser Foundation Research Institute, a Division of Kaiser Permanente Hospitals, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Clinical Research Of Brandon, LLC, Brandon, Florida
  - Access Research Institute, Brooksville, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - I.H.S Health, LLC, Kissimmee, Florida
  - Auzmer Research, Lakeland, Florida
  - Cfagi, Llc, Maitland, Florida
  - Infinite Clinical Research Inc, Miami, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - University of Miami, Miami, Florida
  - MedOne Clinical Research LLC, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Medical Professional Clinical Research Center, Miami, Florida
  - Reliant Medical Research, LLC, Miami, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Ocala GI Research, Ocala, Florida
  - Sarkis Clinical Trials - Parent, Ocala, Florida
  - Endoscopic Research, Inc., Orlando, Florida
  - Arnold Palmer Hospital For Children, Orlando, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - Advanced Research Institute, Inc., Orlando, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Advanced Research Institute, Inc., St. Petersburg, Florida
  - Genesis Clinical Research, Tampa, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Alliance Clinical Research, Tampa, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - One Health Research Clinic Atlanta, LLC, Norcross, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Eagle Clinical Research, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - GI Alliance, Glenview, Illinois
  - GI Alliance, Gurnee, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - The University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - University of Louisville Research Foundation, Louisville, Kentucky
  - GI Alliance - Baton Rouge, Baton Rouge, Louisiana
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - NECCR Primacare Research, LLC, Fall River, Massachusetts
  - Lucida Clinical Trials LLC, New Bedford, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Henry Ford Hospital, Sterling Heights, Michigan
  - Gastrointestinal Associates, PA, Flowood, Mississippi
  - Digestive Health Center PA, Ocean Springs, Mississippi
  - BVL Clinical Research, Liberty, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - AIG Digestive Disease Research, Florham Park, New Jersey
  - NY Scientific Corp., Brooklyn, New York
  - Mount Sinai, New York, New York
  - Rochester Clinical Research, Rochester, New York
  - Charlotte Gastroenterology and Hepatology, P.L.L.C, Charlotte, North Carolina
  - Care Access Research Lumberton, Lumberton, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - Wake Forest Baptist, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Gastro Health Research, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Wexner Medical Center, Columbus, Ohio
  - DSI Research LLC, Springboro, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Board of Regents of the University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Columbia Digestive Health Research, Columbia, South Carolina
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Rapid City Medical Center, LLC, Rapid City, South Dakota
  - Gastroenterology Center of the MidSouth PC, Germantown, Tennessee
  - Digestive Health Research, LC, Hermitage, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Central Texas Clinical Research, LLC, Austin, Texas
  - Amel Med LLC, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - Texas Digestive Disease Consultants, Cedar Park, Texas
  - Baylor Scott and White, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Valley Institute of Research, Fort Worth, Texas
  - GI Alliance - Garland, Garland, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Biopharma Informatic, Inc. Research Center, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Gastro Health & Nutrition, Katy, Texas
  - Mt.Olympus Medical Research, Katy, Texas
  - Digestive System Healthcare, Pasadena, Texas
  - LinQ Research, LLC, Pearland, Texas
  - GI Alliance - San Marcos, San Marcos, Texas
  - GI Alliance - Southlake, Southlake, Texas
  - Texas Gastroenterology Associates, Spring, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - GI Alliance - Webster, Webster, Texas
  - Care Access Research LLC, Ogden, Utah
  - University of Utah, Salt Lake City, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Gastroenterology Consultants and Endoscopy Center of Southwest Virginia, Roanoke, Virginia
  - TPMG Clinical Research Williamsburg, Williamsburg, Virginia
  - University of Washington, Seattle, Washington
  - The Vancouver Clinic, Vancouver, Washington
- Argentina (8):
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Hospital Privado Centro Medico de Cordoba S.A, Córdoba, Córdoba Province
  - Centro de Investigacion CICE, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - CEMIC, Buenos Aires
  - STAT Research S.A., Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
- Australia (13):
  - Blacktown Hospital, Blacktown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Coral Sea Clinical Research Institute, North Mackay, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (5):
  - LKH - Universitaetsklinikum Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - KH der Barmherzigen Brüder St.Veit an der Glan, Sankt Veit an der Glan
- Belgium (11):
  - GZA Ziekenhuizen, Antwerp
  - AZ Klina, Brasschaat
  - C. H. U. St-Pierre, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - AZ Maria Middelares, Ghent
  - AZ Sint-Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - Clinique CHC MontLégia, Liège
  - AZ Delta, Roeselare
  - CHU UCL Namur, Yvoir
- Brazil (12):
  - Hospital Aliança, Salvador, Estado de Bahia
  - L2IP - Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - CDC - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Instituto de Pesquisas em Saúde - Fundação Universidade de Caxias do Sul (IPS/FUCS), Caxias do Sul, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - CECIP - Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Pesquisare Saúde, Santo André, São Paulo
  - Praxis Pesquisa Médica, Santo André, São Paulo
  - Irmandade da Santa Casa da Misericórdia de Santos, Santos, São Paulo
  - Hepatogastro, São Paulo, São Paulo
- Bulgaria (6):
  - Medical center Medconsult Pleven OOD, Pleven
  - DCC "Alexandrovska", EOOD, Sofia
  - UMHATEM 'N.I. Pirogov', EAD, Sofia
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
  - ACIBADEM CityClinic Oncological center, Sofia
  - MC Medica Plus, Veliko Tarnovo
- Canada (6):
  - Gastroenterology and Internal Medicine Research Institute (GIRI), Edmonton, Alberta
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - London Health Sciences Centre (LHSC) - Victoria Hospital, London, Ontario
  - Scott Shulman Medicine Professional Corporation, North Bay, Ontario
  - Toronto Immune & Digestive Health Institute, North York, Ontario
  - Montreal General Hospital, Montreal, Quebec
- China (34):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The 900th Hospital of The Chinese People's Liberation Army Joint Logistics Support Force, Fuzhou, Fujian
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangzhou
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The 2nd Xiangya Hospital of Central South University, Changsha, Hu'nan
  - The First Affiliated Hospital of University of South China, Hengyang, Hu'nan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Renmin Hospital, Wuhan University, Wuhan, Hubei
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Jiangxi Gannan Medical College Affiliated 1 st Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Hua Xiang branch hospital, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Taian City Central Hospital, Tai’an, Shandong
  - Renji Hospital Shanghai Jiaotong University School of Medicine - West Branch, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Tianjin Union Medical Center, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yun'nan
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Croatia (3):
  - General Hospital "Dr.Tomislav Bardek" Koprivnica, Koprivnica
  - Clinical Hospital Centre Osijek, Osijek
  - University hospital centre Zagreb, Zagreb
- Czechia (8):
  - CCR Brno, s.r.o., Brno
  - SurGal Clinic s.r.o., Brno
  - Hepato-Gastroenterologie HK s.r.o., Hradec Králové
  - PreventaMed s.r.o., Olomouc
  - CCR Ostrava s.r.o., Ostrava
  - Fakultni nemocnice Ostrava, Ostrava
  - Institut klinicke a experimentalni mediciny, Prague
  - Nemocnice Slany, Slaný
- France (24):
  - CHU Nice - Hôpital de l'Archet 2, Nice, Alpes Maritimes
  - CHU Reims - Hôpital Robert Debré, Reims, Ardennes
  - Hôpital Nord - CHU Marseille, Marseille, Bouches-du-Rhône
  - CHU Caen - Hôpital de la Côte de Nacre, Caen, Calvados
  - CHU Dijon - Hôpital Bocage Central, Dijon, Cote dÝOr
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac, Gironde
  - Hopital Rangueil, Toulouse, Haute Garonne
  - Institut des MICI, Neuilly, Hauts De Seine
  - Hopital Saint Eloi, Montpellier, Herault
  - CHU Rennes - Hôpital Pontchaillou, Rennes, Ille Et Vilaine
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble, Isère
  - CHU Nantes - Hôtel Dieu, Nantes, Loire Atlantique
  - Universite de Lorraine - Faculte de Medecine - INSERM U954, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - CHU Lille - Hôpital Claude Huriez, Lille, Nord
  - CHU Saint Etienne - Hôpital Nord, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - CHU Clermont Ferrand - Hopital d'Estaing, Clermont-Ferrand, Puy De Dome
  - Centre Hospitalier de Pau - Hôpital François Mitterrand, Pau, Pyrenees Atlantiques
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - CHU Amiens - Hopital Sud, Amiens, Somme
  - Hôpital Henri Mondor, Créteil, Val De Marne
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon, Vendée
  - Hôpital Saint-Louis, Paris
- Germany (18):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Praxis fuer Gasroenterologie Prof. Dr. med Robert Ehehalt, Heidelberg, Baden-Wurttemberg
  - Medius Klinik Nuertingen, Nürtingen, Baden-Wurttemberg
  - Siloah St. Trudpert Klinikum, Pforzheim, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - LMU-Campus Grosshadern, Munich, Bavaria
  - Universitaetsklinikum Frankfurt Goethe-Universitaet, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - INLUGA im Haus der Gesundheit, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig-Holstein
  - Charité - Campus Charité Mitte, Berlin
  - Gastroenterologie Berlin Karlshorst, Berlin
  - Charité - Campus Benjamin Franklin, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Hamburgisches Forschungsinstitut fure Chronische Darmerkrankungen, Hamburg
- Greece (4):
  - General Hospital of Athens "Evangelismos", Athens
  - Corfu General Hospital "St. Eirini", Corfu
  - University General Hospital of Heraklion, Heraklion
  - General Hospital of Thessaloniki "Hippokration", Thessaloniki
- Hungary (6):
  - Bekes Varmegyei Kozponti Korhaz, Békéscsaba
  - Clinexpert Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - Clinfan Szolgaltato Kft., Szekszárd
- India (33):
  - Origin Hospital, Hyderabad, Andhra Pradesh
  - Yashoda Super Speciality Hospital, Hyderabad, Andhra Pradesh
  - Gandhi Hospital, Secunderabad, Andhra Pradesh
  - Navneet Memorial Hospital 'Sushrusha', Ahmedabad, Gujarat
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Gujarat Hospital, Surat, Gujarat
  - Unity Hospital ICU and Trauma, Surat, Gujarat
  - Isha Multispeciality Hospital, Vadodara, Gujarat
  - Fortis Memorial Research Institute, Gurgaon, Haryana
  - M. S. Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - K.L.E. Society's Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagāve, Karnataka
  - Vinaya Hospital and Research Center, Mangalore, Karnataka
  - Lakeshore Hospital and Research Centre Ltd., Kochi, Kerala
  - Amrita Institute Of Medical Sciences and Research Centre, Kochi, Kerala
  - King Edward Memorial Hospital Research Centre, Mumbai, Maharashtra
  - Lokmanya Tilak Municipal General Hospital & Medical College, Mumbai, Maharashtra
  - Kingsway Hospital, Nagpur, Maharashtra
  - Midas Multispeciality Hospital Pvt Ltd, Nagpur, Maharashtra
  - Chopda Medicare & Research Centre, Nashik, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Sahyadri Specialty Hospital, Pune, Maharashtra
  - Datta Meghe Institute of Medical Sciences (Deemed University), Wardha, Maharashtra
  - Fortis Escorts Heart Institute and Research Centre, New Delhi, National Capital Territory of Delhi
  - Maharaja Agrasen Hospital, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - S. R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - SRM Institutes for Medical Sciences, Chennai, Tamil Nadu
  - Chhatrapati Shahuji Maharaj (CSM) Medical University, Lucknow, Uttar Pradesh
  - Nil Ratan Sircar Medical College, Kolkata, West Bengal
  - Institute of Post Graduate Medical Education And Research, Kolkata, West Bengal
  - Postgraduate Institute of Medical Education and Research, Chandigarh
- Ireland (5):
  - Midland Regional Hospital, Mullingar, Westmeath
  - Connolly Hospital, Dublin
  - St Vincents University Hospital, Dublin
  - Portiuncula Hospital, Galway
  - Our Lady of Lourdes, Louth
- Israel (10):
  - HaEmek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center KMC Institute of Gastroenterology and Liver Diseases, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (22):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Ospedale di Circolo, Rho, Milano
  - Ospedale San Raffaele, Rozzano, Milano
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese, Milano
  - Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Azienda Ospedaliera Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Azienda Ospedaliera Giuseppe Brotzu, Cagliari
  - Presidio Ospedaliero Garibaldi Nesima, Catania
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana (Presidio di Cisanello), Pisa
  - Università Campus Bio-Medico di Roma, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
  - Ospedale San Bortolo di Vicenza, Vicenza
- Japan (48):
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Kokikai Tsujinaka Hospital Kashiwanoha, Kashiwa-shi, Chiba
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Aso Co.,Ltd Iizuka Hospital, Iizuka-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Our Lady of the Snow St. Mary's Hospital, Kurume-shi, Fukuoka
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ota-shi, Gunma
  - NHO Fukuyama Medical Center, Fukuyama-shi, Hiroshima
  - JA-Hiroshima General Hospital, Hatsukaichi-shi, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - NHO Kure Medical Center and Chugoku Cancer Center, Kure-shi, Hiroshima
  - Asahikawa Medical University Hospital, Asahikawa-shi, Hokkaido
  - JCHO Hokkaido Hospital, Sapporo, Hokkaido
  - Aoyama Clinic, Kobe, Hyōgo
  - NHO Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Jiaikai Izuro Imamura Hospital, Kagoshima, Kagoshima-ken
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima, Kagoshima-ken
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Gokeikai Ofuna Chuo Hospital, Kamakura-shi, Kanagawa
  - Kawasaki Municipal Hospital, Kawasaki-shi, Kanagawa
  - Keijinkai Matsushima Hospital, Yokohama, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Kaiseikai Hattori Clinic, Kumamoto, Kumamoto
  - Mie University Hospital, Tsu, Mie-ken
  - Nagaoka Red Cross Hospital, Nagaoka-shi, Niigata
  - Saiseikai Niigata Hospital, Niigata, Niigata
  - Ishida Clinic of IBD and Gastroenterology, Ōita, Oita Prefecture
  - Okayama University Hospital, Okayama, Okayama-ken
  - NHO Okayama Medical Center, Okayama, Okayama-ken
  - Keiaikai Nakagami Hospital, Okinawa-shi, Okinawa
  - Shinseikai Sai Gastroenterology, Proctology, Fujiidera-shi, Osaka
  - Kinshukai Infusion Clinic, Osaka, Osaka
  - NHO Osaka National Hospital, Osaka, Osaka
  - JCHO Osaka Hospital, Osaka, Osaka
  - Saga-Ken Medical Centre Koseikan, Saga, Saga-ken
  - Saga University Hospital, Saga, Saga-ken
  - NHO Ureshino Medical Center, Ureshino-shi, Saga-ken
  - Kumagaya General Hospital, Kumagaya-shi, Saitama
  - Matsuaikai Matsuda Hospital, Hamamatsu, Shizuoka
  - Tokyo Medical and Dental University Hospital, Bunkyō City, Tokyo-To
  - Showa University Koto Toyosu Hospital, Kōtoku, Tokyo-To
  - Kitasato University Kitasato Institute Hospital, Minatoku, Tokyo-To
  - JCHO Tokyo Yamate Medical Center, Shinjuku-Ku, Tokyo-To
  - Tokyo Metropolitan Bokutoh Hospital, Sumida-ku, Tokyo-To
  - NHO Mito Medical Center, Ibaraki
- Lithuania (3):
  - Lithuanian University of Health Sciences Kaunas Hospital, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Klaipeda University Hospital branch "Seamen's Hospital", Klaipėda
- Mexico (6):
  - Consultorio Medico, InvesclinicMX, Irapuato, Guanajuato
  - Accelerium S de RL de CV, Monterrey, Nuevo León
  - Inspirepharma S. de R.L. de C.V., Monterrey, Nuevo León
  - Christus Muguerza Sur S.A. de C.V., Monterrey, Nuevo León
  - FAICIC S. de R.L. de C.V., Veracruz
  - Sociedad de Metabolismo y Corazon S.C, Veracruz
- Netherlands (7):
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Zuyderland Medisch Centrum - Sittard-Geleen, Geleen
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - ETZ Elisabeth, Tilburg
  - Bernhoven Uden, Uden
  - UMC Utrecht, Utrecht
- New Zealand (4):
  - Christchurch Hospital NZ, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Tauranga Hospital, Tauranga
- Poland (31):
  - Przychodnia Specjalistyczna Insula, Bełchatów
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Trialmed CRS, Kalisz
  - Polimedica Centrum Badań, Profilaktyki I Leczenia, Kielce
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Centrum Medyczne Plejady, Krakow
  - NZOZ Centrum Medyczne ProMiMed, Krakow
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - AMICARE spółka z ograniczoną odpowiedzialnością spółka komandytowa, Lodz
  - 1 Wojskowy Szpital Kliniczny z Polikliniką SPZOZ w Lublinie, Lublin
  - ALLMEDICA sp. z o. o., Nowy Targ
  - Wojewodzki Specjalistyczny Szpital w Olsztynie, Olsztyn
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - Medicome Sp. z o.o., Oświęcim
  - SOLUMED Centrum Medyczne, Poznan
  - NSZOZ Termedica - Centrum Badan Klinicznych, Poznan
  - Twoja Przychodnia PCM, Poznan
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Kiepury Clinic MAŁGORZATA JARNOT SPECJALISTYCZNA PRAKTYKA GINEKOLOGICZNO-POŁOŻNICZA, Sosnowiec
  - KO-MED Centra Kliniczne Staszow, Staszów
  - DC-MED, Swidnica
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne Sp. z o. o., Szczecin
  - CenterMed Sp. z o.o., Tarnów
  - Centrum Zdrowia MDM, Warsaw
  - NZOZ VIVAMED Jadwiga Miecz, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - Ars-Medica S.C Rybak Maria, Rybak Zbigniew, Wroclaw
  - ETG Zamosc, Zamość
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Lecznej, Łęczna
- Portugal (6):
  - Hospital de Braga, Braga
  - Hospital da Senhora da Oliveira Guimarães, Guimarães
  - Hospital da Luz, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E - Hospital de São Sebastião, Santa Maria da Feira
  - Centro Hospitalar do Alto Minho - Unidade Local de Saúde do Alto Minho, EPE, Viana do Castelo
- Romania (8):
  - SC Centrul Medical Medicum SRL, Specialitatea Gastroenterologie, Bucharest
  - Spitalul de Oncologie Monza, Bucharest
  - S.C Delta Health Care S.R.L, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - Centrul Medical Renasterea Craiova, Craiova
  - S.C Pelican Impex S.R.L, Oradea
  - S.C Centrul Medical Valahia S.R.L, Ploieşti
- Serbia (6):
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Clinical Hospital Center "Bezanijska kosa, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - General Hospital Subotica, Subotica
  - General Hospital "Djordje Joanovic", Zrenjanin
- Slovakia (8):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Cliniq s.r.o., Bratislava
  - Endomed, s.r.o., Košice
  - KM Management spol. s r.o., Nitra
  - Fakultna nemocnica Nitra, Nitra
  - Gastro I, s.r.o., Prešov
  - Gastro LM s.r.o., Prešov
  - Accout Center s.r.o., Šahy
- South Korea (20):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Yeungnam University Hospital, Daegu, Gyeongsangbuk-do
  - Korea University Ansan Hospital, Ansan-si, North Chungcheong
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
- Spain (18):
  - Hospital Universitario Reina Sofia, Córdoba, Cordoba
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, La Coruña
  - Clinica Gaias - Santiago, Santiago de Compostela, La Coruña
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Centro Medico Teknon, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital General Juan Ramon Jimenez, Huelva
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Montecelo, Pontevedra
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (4):
  - Clarunis - Universitäres Bauchzentrum Basel, Basel
  - Inselspital - Universitaetsspital Bern, Bern
  - Intesto Gastroenterologische Praxis, Crohn-Colitis-Zentrum Bern, Bern
  - Universitaetsspital Zuerich, Zurich
- Turkey (Türkiye) (9):
  - Gazi University Medical Faculty, Ankara
  - Antalya Training and Research Hospital, Antalya
  - Koc University Hospital, Istanbul
  - Medicana Kadikoy Hospital, Istanbul
  - Acibadem Kozyatagi Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Inonu University Gastroenterology, Malatya
  - Mersin University Medical Faculty, Mersin
- United Kingdom (10):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - Guy's Hospital, London, Greater London
  - King's College Hospital, London, Greater London
  - Hammersmith Hospital, London, Greater London
  - Bury Care Organisation, Bury, Greater Manchester
  - St Mark's Hospital, Harrow, Middlesex
  - Yeovil District Hospital, Yeovil, Somerset
  - Huddersfield Royal Infirmary, Huddersfield, West Yorkshire
  - The Ulster Hospital, Belfast